CLINICAL TRIAL: NCT01896700
Title: Methylphenidate to Improve Balance and Walking in MS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Cameron, Neurologist, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3055
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; postural balance; walking
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Intervention: An escalating dose of methylphenidate taken by mouth: 20mg for 2 weeks, 40mg for 2 weeks, 60mg for 2 weeks. All doses divided twice/day.
  Other name: Ritalin
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Placebo pill, bid for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Escalating dose of methylphenidate, 20mg, 40mg, 60mg/day, for 2 weeks each
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo — Escalating matched dose of placebo
  Arms: Placebo

SUMMARY:
Methylphenidate is an amphetamine-like psychomotor stimulant drug currently approved for the treatment of attention-deficit hyperactivity disorder (ADHD), postural orthostasis tachycardia syndrome and narcolepsy. It is also often prescribed off label to people with MS to improve fatigue. It is proposed that methylphenidate may also improve imbalance and walking deficits in MS by improving concentration and central integration, one of the primary mechanisms thought to underlie imbalance and walking deficits in MS.

DETAILED DESCRIPTION:
The proposed pilot study will examine the effects of methylphenidate on imbalance and walking in 24 subjects with MS and imbalance. The subjects will be randomly assigned to receive either an escalating does of methylphenidate, 20mg, 40mg or 60mg, divided into two doses each day, or matched placebo for 2 weeks at each dose. If a subject does not tolerate dose escalation they will be instructed to discontinue use of the drug. The maximum safely tolerated dose for each subject will be noted. Changes from baseline in subject's walking speed, balance, vestibular function, cognitive function, and fatigue will be assessed at each dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65
* Able to walk at least 100m without an aide or with unilateral assistance
* Poor static balance, specifically prolonged APR latencies (≥ 1 standard deviation (SD) > mean for healthy people in this age range), OR
* Reduced balance-related activity (ABC scores ≤ 85%)
* Walking difficulties, specifically T25FW > 6 seconds, OR reduced self perceived walking (MSWS-12 scores ≥ 50/60)

Exclusion Criteria:

* Currently taking methylphenidate, modafinil, or armodafinil.(any within the last 2 weeks)
* Cause(s) of imbalance other than MS
* Systolic pressure consistently greater than 150 mm Hg or diastolic pressure consistently greater than 90 mm Hg
* Contraindications to methylphenidate (Anxiety, tension, agitation, thyrotoxicosis, tachyarrhythmias, severe angina pectoris or glaucoma, hypersensitivity to methylphenidate, motor tics or a family history or diagnosis of Tourette's syndrome, seizures, severe or poorly controlled hypertension, treatment with monoamine oxidase inhibitors currently or within the last 14 days, current use of guanethidine, pressors, coumarin anticoagulants, anticonvulsants, phenylbutazone, or tricyclic antidepressants, history of drug abuse or alcoholism)
* Pregnancy or breastfeeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cameron, PT, MD, Principal Investigator — Portland VA Medical Center
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 people with MS and imbalance from the MS clinics in the Portland, OR metropolitan area were enrolled into this study between September 2013 and March 2016 .
Groups:
- Methylphenidate: Intervention: An escalating dose of methylphenidate taken by mouth: 20mg for 2 weeks, 40mg for 2 weeks, 60mg for 2 weeks. All doses divided twice/day.
  Other name: Ritalin
  Methylphenidate: Escalating dose of methylphenidate, 20mg, 40mg, 60mg/day, for 2 weeks each
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 12 | 12
Completed | 8 | 6
Not Completed | 4 | 6
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (7.9) | 51.7 (8.7) | 49.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Timed Up and Go (TUG) Test Time at 6 Weeks
Description: The primary outcome of this study will be the difference between mean change in TUG time between methylphenidate and placebo treated subjects at 6 weeks. Mean changes will be compared for active and placebo treated subjects using Bayesian analysis.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: change in seconds from basline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 8 | 6
change in seconds from basline | -0.7 (0.5) | -1.3 (0.2)

2. Secondary Outcome: Change From Baseline in Automatic Postural Response (APR) Latency at 6 Weeks
Description: Mean changes in APR latency at 6 weeks will be compared for active and placebo treated subjects using Bayesian analysis.
Time Frame: 6 weeks
Population: Population discrepancy: One participant in the intervention group and two participants in the placebo group contributed unusable APR data; due to their balance deficits, the machine could not get an accurate reading for this test. One participant in the intervention group declined this test. These four participants were not included in analysis.
Measure: Mean (Standard Error); unit: change in milliseconds from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 6 | 4
change in milliseconds from baseline | -9.2 (2.2) | -5.3 (1.8)

3. Secondary Outcome: Change From Baseline in Timed 25 Foot Walk (T25FW) at 6 Weeks
Description: Mean changes in Timed 25 Foot Walk (T25FW) at 6 weeks will be compared for active and placebo treated subjects using Bayesian analysis.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: change in seconds from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 8 | 6
change in seconds from baseline | -0.3 (0.7) | -0.6 (0.2)

4. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Assessment Questionnaire Score at 6 Weeks
Description: Mean changes in the score attained on the Pittsburgh Sleep Quality Assessment Questionnaire at 6 weeks will be compared for active and placebo treated subjects using Bayesian analysis. Scale ranges from 0-21 points, with higher numbers indicating poorer sleep quality.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: change in score from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 8 | 6
change in score from baseline | 0.3 (0.9) | -0.3 (0.7)

5. Secondary Outcome: Change From Baseline in Modified Fatigue Index Scale Score at 6 Weeks
Description: Mean changes in the score attached on the Modified Fatigue Index Scale at 6 weeks will be compared for active and placebo treated subjects using Bayesian analysis. Scale ranges from 0-84 points, with higher scores indicating greater fatigue.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: change in score from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 8 | 6
change in score from baseline | -3.8 (3.5) | -9.8 (4.4)

6. Secondary Outcome: Change From Baseline in Vestibular-Ocular Reflex (VOR) Gain at 6 Weeks
Description: The most common rotary chair testing is a battery of subtests, each at a specific rate (Hz) of chair rotation from side to side. The participant is secured in the chair in total darkness while the eyes are monitored by infrared cameras. We completed tests from 0.04 to 0.64 Hz to assess the vestibular system across a range of head movements. The chair and participant's head move together while the cameras track the velocity of the eyes; eye velocity reveals how the vestibular system responds to head velocity. VOR gain is the ratio of average chair (i.e. head) velocity to average eye velocity, and is represented on a unitless scale from 0 to 1. VOR gain close to 1 indicates that eye velocity is nearly equal and opposite to head velocity. While there are normative ranges for VOR gain, we are most interested in is change in mean gain (6-week tests minus baseline tests) for the active and placebo groups.
Time Frame: 6 weeks
Population: Explanation of population discrepancy: One participant in the active group declined this test, so was not analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 7 | 6
ratio
  VOR Gain at 0.04 Hz | -0.0107 (0.0868) | -0.0229 (0.0521)
  VOR Gain at 0.08 Hz | -0.0061 (0.0759) | -0.283 (0.0340)
  VOR Gain at 0.16 Hz | -0.0151 (0.0949) | 0.0871 (0.0702)
  VOR Gain at 0.32 Hz | -0.0422 (0.1154) | 0.0322 (0.0680)
  VOR Gain at 0.64 Hz | 0.0221 (0.0894) | 0.0151 (0.0614)

7. Secondary Outcome: Change From Baseline in Vestibular Ocular Reflex (VOR) Asymmetry (Percentage Asymmetric) at 6 Weeks
Description: Mean changes in VOR asymmetry, which is a measure of the strength of the eye responses in one direction compared with the other as measured by rotary chair testing at 6 weeks, will be compared for active and placebo treated subjects using t-tests, or other appropriate statistical analyses. A range of frequencies was tested from 0.04 Hz to 0.64 Hz, as is standard for rotary chair testing. The range of frequencies (i.e. chair speeds) assesses the vestibular system across a range of head movements. This helps to identify abnormality, which may manifest at different frequencies of movement. The measurement outcomes for rotary chair testing are gain, phase and asymmetry of the eye movements.
Time Frame: 6 weeks
Population: Explanation of population discrepancy: One participant in the active group declined this test, so was not analyzed.
Measure: Mean (Standard Deviation); unit: change in % of asymmetry from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 7 | 6
change in % of asymmetry from baseline
  VOR Asymmetry at 0.04 Hz | 0.9927 (5.6664) | -1.7291 (2.3367)
  VOR Asymmetry at 0.08 Hz | -0.0572 (5.6678) | -6.5209 (1.9883)
  VOR Asymmetry at 0.16 Hz | 2.5833 (3.1565) | -5.2852 (4.9239)
  VOR Asymmetry at 0.32 Hz | 1.9157 (5.1153) | -4.1203 (5.4695)
  VOR Asymmetry at 0.64 Hz | 0.3104 (4.0893) | -1.5111 (3.7015)

8. Secondary Outcome: Change From Baseline in Vestibular Ocular Reflex (VOR) Phase (in Degrees) at 6 Weeks
Description: Mean changes in VOR phase, which is a measure of the timing (in degrees) of the eye movements relative to the chair movement, as measured by rotary chair testing at 6 weeks, will be compared for active and placebo treated subjects using t-tests, or other appropriate statistical analyses. A range of frequencies was tested from 0.04 Hz to 0.64 Hz, as is standard for rotary chair testing. The range of frequencies (i.e. chair speeds) assesses the vestibular system across a range of head movements. This helps to identify abnormality, which may manifest at different frequencies of movement. The measurement outcomes for rotary chair testing are gain, phase and asymmetry of the eye movements.
Time Frame: 6 weeks
Population: Explanation of population discrepancy: One participant in the active group declined this test, so was not analyzed.
Measure: Mean (Standard Deviation); unit: change in degrees from baseline
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 7 | 6
change in degrees from baseline
  VOR Phase at 0.04 Hz | 2.2790 (5.2622) | 1.9535 (4.2274)
  VOR Phase at 0.08 Hz | 1.8914 (4.2548) | -1.4716 (2.5754)
  VOR Phase at 0.16 Hz | 0.9449 (2.2400) | -0.3342 (3.6845)
  VOR Phase at 0.32 Hz | -1.3564 (7.0617) | 0.5981 (3.6808)
  VOR Phase at 0.64 Hz | -2.7082 (3.6010) | 0.2833 (1.7800)

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events during the 6 weeks of their participation in the study.
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=12) | Placebo (N=12)
Elevated blood pressure (Vascular disorders) | 1 | 3
Elevated heart rate (Cardiac disorders) | 1 | 0
Chest pain/tightness (General disorders) | 1 | 0
Headache (General disorders) | 2 | 2
Insomnia (General disorders) | 6 | 4
Nightmares (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Stomach ache/indigestion (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal cramping (General disorders) | 0 | 1
Reduced appetite (Metabolism and nutrition disorders) | 1 | 0
Agitation (General disorders) | 2 | 0
Irritation (General disorders) | 1 | 0
Emotional detachment (General disorders) | 1 | 0
Spasms of limbs (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Itchiness (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Tingling sensation (General disorders) | 1 | 0
Increased body heat (General disorders) | 1 | 1
Coughing/sneezing/respiratory effects (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dry mouth (General disorders) | 2 | 0
Dizziness (General disorders) | 1 | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat/ear infection (Infections and infestations) | 1 | 0
Reduced balance (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3
Car accident (Injury, poisoning and procedural complications) | 1 | 0
MS relapse (Nervous system disorders) | 1 | 0
Family emergency (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes